CLINICAL TRIAL: NCT02394067
Title: Magnetic Resonance Venography Pre- and Post-Treatment in Patients With Idiopathic Intracranial Hypertension
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 20150217
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2022-10

CONDITIONS: Pseudotumor Cerebri
MeSH Terms: conditions — Pseudotumor Cerebri | interventions — Postmortem Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Idiopathic Intracranial Hypertension: All participants of our study will be in this arm. These will be patients with a diagnosis of IIH. These patients will be followed throughout their standard of care treatment, with neuro-radiological imaging.
  Interventions: Other: Radiological Imaging

INTERVENTIONS:
Other: Radiological Imaging — magnetic resonance imaging and magnetic resonance venography scans

SUMMARY:
This prospective study will use magnetic resonance imaging of patients with Idiopathic Intracranial Hypertension (IIH), to determine if the common radiological finding of transverse venous sinus stenosis can be reversed with standard of care medical treatment of IIH.

DETAILED DESCRIPTION:
Patients with suspected Idiopathic Intracranial Hypertension (IIH) will be recruited and undergo an ophthalmologic investigation, and a lumbar puncture, both of which are necessary for diagnosis of IIH. MRI is done as a standard of care to rule out other etiologies of raised intracranial pressure. Our patients will require four MRI/MRVs. The first MRI/MRV is standard of care scan. The second MRI/MRV will be on the day of the lumber puncture, immediately following the procedure. The third MRI/MRV will take place when significant reduction of clinical papilledema has taken place (about 3-6 months), and a forth MRI will take place one year after the initial presentation or with symptom resolution, whichever comes first. Radiological findings will be compared at all stages to determine if transverse venous sinus stenosis can be reversed with standard of care medical treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients with a diagnosis of IIH, where other intracranial pathology has been ruled out, can participate.

Exclusion Criteria:

(1)Patients who have a contraindication or are unable to undergo magnetic resonance imaging. (2)Patients who are found to have intracranial pathology to explain elevated intracranial pressure. (3)Patients with allergies to gadolinium-containing agents.(4)Patients with elevated creatinine above normal laboratory values.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from the neuro-ophthalmology service at the Queen Elizabeth II Health Center. Neuro-ophthalmology service in Nova Scotia sees approximately 20 new diagnoses of IIH per year.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Transverse venous sinus stenosis (combined conduit score, and measure of transverse venous sinus stenosis, for each MRI/MRV) | 4 MRI/MRV's performed within a year of diagnosis
  The main outcome measure will be a combined conduit score, and measure of transverse venous sinus stenosis, for each MRI/MRV.

CONTACTS AND LOCATIONS:
Overall Officials: Jai Shankar, MD, Principal Investigator — Capital Health, Canada
Locations (1):
- CapitalDHACanada, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No